CLINICAL TRIAL: NCT07321821
Title: The Effect of Fermented Garlic Lettuce Powder on Cognitive Function in Adults With Mild Cognitive Impairment: An Investigator-Initiated, Randomized, Assessor-Blinded, Parallel-Group, Controlled, Single-Center Study
Brief Title: Fermented Garlic Lettuce Powder and Cognitive Function in Adults With Mild Cognitive Impairment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Yong-il Shin, Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11-2024-061
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Mild Cognitive Impairment (MCI)
Keywords: Fermented Garlic Lettuce Powder; Mild Cognitive Impairment; Psychological Outcome; Randomized Controlled Trial
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Participants with mild cognitive impairment (K-MoCA scores 16-23) will be randomly assigned to either the intervention group receiving fermented garlic lettuce powder daily for 2 months or to a control group. Cognitive and psychological outcomes will be assessed at baseline and at the end of the 2-month intervention. Outcome assessors will be blinded to group allocation, and the study will be conducted as a single-center, investigator-initiated, parallel-group, randomized controlled trial.
Who Masked: Outcomes Assessor
Masking Description: except for one assessor who will have access to group assignments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fermented Garlic Lettuce Powder (Experimental): Participants receive fermented garlic lettuce powder, administered orally as three tablets per day for 2 months (total of 180 tablets).
  Interventions: Dietary Supplement: Garlic Lettuce Fermented Powder
- Placebo Tablet (Placebo Comparator): Participants take 1 placebo tablet daily for 2 months, totaling 60 tablets
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Garlic Lettuce Fermented Powder — The Garlic Lettuce Fermented Powder tablets (intervention group) are taken 3 tablets daily for 2 months, totaling 180 tablets
  Arms: Fermented Garlic Lettuce Powder
Other: Placebo — Participants take 1 placebo tablet daily for 2 months, totaling 60 tablets
  Arms: Placebo Tablet

SUMMARY:
"This study aims to investigate the cognitive and psychological changes in adults with mild cognitive impairment (K-MoCA scores between 16 and 23) following daily consumption of fermented garlic lettuce powder for 2 months

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 years or older with K-MoCA scores between 16 and 23.
* Individuals with sufficient vision and hearing to participate in the study without difficulty.
* Participants who are currently taking medications or receiving treatments that may affect cognition and are able to maintain the same dosage and regimen throughout the study period.
* Individuals who voluntarily agree to participate in the study and provide written informed consent.

Exclusion Criteria:

* Individuals who have undergone vascular-related surgery within the past 6 months or gastrointestinal surgery that may affect absorption of the study product (excluding simple appendectomy or hernia repair).
* Individuals with a clinically significant history of hypersensitivity to medications or dietary supplements.
* Individuals with a history of alcohol or drug abuse.
* Individuals unable to communicate effectively.
* Individuals who have participated in more than two dietary supplement studies or clinical trials within the current year, or within the past 6 months.
* Individuals deemed unable to participate safely or effectively in the study by the investigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-09-19 (Actual); Primary Completion 2026-01-21 (Estimated); Study Completion 2026-01-21 (Estimated)

PRIMARY OUTCOMES:
K-MoCA | Assessments are performed at baseline and at 2 months.
  The Korean version of the Montreal Cognitive Assessment (K-MoCA) is a cognitive screening tool with scores ranging from 0 to 30, with higher scores indicating better cognitive function. The outcome measure is the change in K-MoCA score.

SECONDARY OUTCOMES:
SVLT | Assessments are performed at baseline and at 2 months.
  The Seoul Verbal Learning Test (SVLT) is a neuropsychological assessment tool used to evaluate verbal memory performance. Scores range from 0 to 36, with higher scores indicating better memory function.
KCWS | Assessments are performed at baseline and at 2 months.
  The Korean Color-Word Stroop Test (KCWS) is a neuropsychological assessment used to evaluate executive function and cognitive control. Performance is measured by the number of correct responses within 1- and 2-minute intervals, with higher scores indicating better cognitive function.
RCFT | Assessments are performed at baseline and at 2 months.
  The Rey Complex Figure Test (RCFT) is a neuropsychological assessment used to evaluate visuospatial constructional ability and visual memory. Scores range from 0 to 36, with higher scores indicating better memory performance.
DST | Assessments are performed at baseline and at 2 months.
  The Digit Span Test (DST) is a neuropsychological assessment used to evaluate attention and working memory. Scores range from 0 to 24, with higher scores indicating better concentration and attention.
COWAT | Assessments are performed at baseline and at 2 months.
  The Controlled Oral Word Association Test (COWAT) is a neuropsychological assessment used to evaluate verbal fluency and executive function. Scores range from 0 to 27, with higher scores indicating better verbal fluency, executive function, attention, and problem-solving abilities.
BDI | Assessments are performed at baseline and at 2 months.
  The Beck Depression Inventory (BDI) is a self-report questionnaire used to assess the severity of depressive symptoms. Each item is scored from 0 to 3, with total scores ranging from 0 to 63, where higher scores indicate more severe depressive symptoms.
EQ-5D | Assessments are performed at baseline and at 2 months.
  The EuroQol-5 Dimension (EQ-5D) is a standardized instrument for measuring health-related quality of life. Scores range from 0 to 100, with lower scores indicating better perceived health status and higher scores reflecting more severe health problems.
MFS | Assessments are performed at baseline and at 2 months.
  The Multidimensional Fatigue Scale (MFS) is a self-report questionnaire used to assess fatigue across multiple dimensions. Each dimension is rated from 0 to 20, with a total score ranging from 0 to 100. Lower scores indicate less fatigue, while higher scores reflect more severe fatigue.
PWI-SF | Assessments are performed at baseline and at 2 months.
  The Psychological Well-Being Index-Short Form (PWI-SF) is a self-report questionnaire used to assess psychological well-being. Each dimension is rated from 0 to 20, with total scores ranging from 0 to 54, where higher scores indicate better psychological well-being, life satisfaction, and emotional stability.
LSEQ | Assessments are performed at baseline and at 2 months.
  The Leeds Sleep Evaluation Questionnaire (LSEQ) is a self-report instrument used to assess subjective sleep quality. Scores are based on a scale from 0 to 100, with higher scores indicating better sleep quality and lower scores reflecting greater sleep disturbance.

CONTACTS AND LOCATIONS:
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No